CLINICAL TRIAL: NCT06473181
Title: The Impact Of Core Stability Exercises On Standing , Functional Balance And Gait In Diplegic Cerebral Palsy Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, nancy mohamed eid metwaly shaban, Clinical professor, Kafrelsheikh University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KFSIRB200-162
Record Dates: First submitted 2024-05-24; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Diplegic Cerebral Palsy With Spasticity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Core stability exercises that is part of physiotherapy rehabilitation (Other): Physical therapy including core stability exercises and improving developmental milestones to improve children development
  Interventions: Other: Core stability exercises

INTERVENTIONS:
Other: Core stability exercises — Exercises applied to trunk , pelvis and abdomen to improve ability to stand , walk and balance.

SUMMARY:
The term of "core stability" explains the capacity to control the position and movement of the central portion of the body. Core stability training targets the muscles deep within the abdomen that attach to the spine, pelvis and shoulders, that help in the preservation of proper posture and provide the basis for movements of extremities in a coordinated manner. The aim of core stability training is to achieve the optimal physical ability tom the normal state of the spine in daily activities, in addition to developing the endurance and coordination of these core stability muscles.The Core stability may help to improve dynamic balance and muscle coordination between lower and upper extremities, as well as reducing injury risk and muscle imbalances . Core stability exercises have a positive effect on reducing pain, activating deep abdominal muscles, elevating the stability of lumbar spine and improving physical function in patients . The stability of the lumbo-pelvic region is crucial to provide a foundation for movement of the upper and lower extremities, to support loads, and to protect the spinal cord and nerve roots . The core muscles stabilize the spine and trunk during movements such as jumping, running, and throwing .

DETAILED DESCRIPTION:
Cerebral palsy (CP) could be a cluster of disorders that have an effect on the event of movement and posture,inflicting activity limitation, and nonprogressive disturbances that occurred within the developing fetal or child brain.The main therapeutic goals for children with CP are the performance of functional activities and walking.

Children with CP have a limitation with activities due to the existing impairments in independent walking, climbing stairs, running, or walking over uneven surface .Functional limitation of children with CP may have various degrees due to loss of axial control with an imbalance of their movement .Balance has been defined as the elements of postural control that allow a child to safely perform everyday tasks . Poor balance control is one of the most contributing factors for poor gait and reaching movement because the maintenance of stability is critical to all movements . Children with CP have defects in postural mechanisms, including righting and equilibrium reactions, antigravity mechanism, proximal stability, and postural fixation . Diplegia is amongst the most widely recognized clinical subtypes of Cerebral Palsy (CP). It is used when the motor impairment is milder in the upper limbs than the lower limbs. Most children have major weakness in the trunk and hypertonic limbs .Diplegia is characterized by increased muscle tone with difficulty in relaxing. Active movements are slow and stiff with abnormal patterns. Lower limbs are more affected than upper limbs. Head and neck are unaffected but there is weakness and limited rotation of the trunk . Children with CP may experience a range of functional limitations as a result of loss of trunk control and movement imbalance. Balance is defined as the postural control elements which enable a child to safely execute daily tasks.Because maintaining stability is necessary for all movements, low balance control is one of the extreme common causes of unsafe walking or reaching function . So core stability training is preferred to maintain position and movement of body core. Stability training involves the abdomen muscles and pelvic and shoulder muscles, which maintain postural alignment and allow movements of extremities. Postural control is mainly for motion and depends on these muscles for stability and endurance. Components of core stability include strength, endurance, balance,nd the related activity of the back, abdominal, and pelvic muscles . The core muscles act like one block to keep the body stable during static state and with extremity motion . CP children lack the ability to distribute the load, that is, body weight, appropriately during static balance and transfer the body weight adequately from one supporting limb to another during dynamic balance tasks . Children with diplegic CP are characterized by impairment of motor control in the lower extremities more than in the upper extremities.

Statement of the problem This study will be conducted to answer the following research question:Is there any significant effect of core stability exercises on standing , balance and gait in Diplegic cerebral palsy children ? Purpose of the study The purpose of this study is to study the effect of core stability training on standing, balance and gait in spastic diplegic cerebral palsy children.

Significance of the study Spasticity, muscle contraction, bony malformations, loss of selective motor control, and muscle weakness are potential factors that interfere with normal gait patterns in diplegic CP. Recent studies have found that muscle weakness limits motor function in children with CP more than spasticity. Therefore, strengthening weak muscles is es-sential for spasticity management to improve the func-tion of diplegic CP.Balance disorder is a serious problem for children with diplegic CP, and this can make it difficult to achieve and maintain equilibrium. Children with diplegic CP have reduced neuromotor perceptual func-tion, inadequate stance stability in different sensory settings, slow anticipatory response, and inaccurate pre-paratory activation.

The term of "core stability" explains the capacity to control the position and movement of the central portion of the body. Core stability training targets the muscles deep within the abdomen that attach to the spine, pelvis and shoulders, that help in the preservation of proper posture and provide the basis for movements of extremities in a coordinated manner. Spinal stability is essential for the production of movement and relies on the core muscles to acquire sufficient strength, power, and endurance .The core has illustrated by researchers as a "power-house" for initiating limb movement or as a double-walled cylinder or box in which the abdominals act as the front of the house, the paraspinals serve as the back, the diaphragm serves as the roof, and the musculature of the hip girdle and pelvic floor create the 2 basement of the house.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of diplegic CP made by paediatricians or pediatric neurologists
* children spasticity grades must range from 1 to 1+ according to MAS
* age must range from 4 to 10 years
* They Must be in level I or II on the Gross Motor Function Classifcation System (GMFCS)

Exclusion Criteria:

* A permanent deformity (bony or soft tissue contractures)
* visual or auditory defects
* Botox application to the lower extremity in the past 6 months or undergone a previous surgical intervention to ankle and knee
* history of epileptic seizure and any diagnosed cardiac or orthopaedic disability

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Pediatric balance scale | Baseline
  To assess the static balance Pediatric Balance Scale scores are divided into 14 items, scored between 0 to 4. What counts as 0 and 4 will vary from exercise to exercise, but 0 is considered the worst performance, and 4 is the best.
  Retrials are unnecessary if they score a 4 on the first trial. Since each exercise has three trials, the score rating you must tick for each item should be the best of the three trials.
  Some exercises have time and distance requirements. Points will be deducted if they cannot complete the time and distance requirements and require external support or assistance from another person.
  After all the exercises have been performed, you simply need to add up all the score ratings per item to calculate the total test score.
  The maximum score is 56.
Gross motor function classification system | Baseline
  To assess the gross motor function and standing The GMFM is a standardized observational instrument designed and validated to measure change in gross motor function over time in children with cerebral palsy. The scoring key is meant to be a general guideline.
  However, most of the items have specific descriptors for each score. It is imperative that the guidelines contained in the manual be used for scoring each item. SCORING KEY 0 = does not initiate
  1. = initiates
  2. = partially completes
  3. = completes
Modified Ashworth scale | Baseline
  To measure the degree of spasticity to enroll children in the study
  scoring
  0 No increase in tone
  1 slight increase in tone giving a catch when slight increase in muscle tone, manifested by the limb was moved in flexion or extension.
  1+ slight increase in muscle tone, manifested by a catch followed by minimal resistance throughout (ROM )
  2 more marked increase in tone but more marked increased in muscle tone through most limb easily flexed
  3 considerable increase in tone, passive movement difficult
  4 limb rigid in flexion or extension
Weight-Height scale | Baseline
  To measure weight and height to calculate BMI for each patient . The child was wearing a thin layer of clothes to calculate BMI according to the following equation: BMI (Kg/m²)= weight(kg) ÷ height²(m2)

CONTACTS AND LOCATIONS:
Overall Officials: Core stability training In Diplegic Cerebral Palsy, Master, Principal Investigator — Kafr Elsheikh